CLINICAL TRIAL: NCT01513694
Title: Clinical Trial Phase I / II Prospective, Open, Non-randomized for Treatment of Lumbar Intervertebral Degenerative Disc Disease With Posterolateral Instrumented and Autologous Mesenchymal Stem Cells.
Brief Title: Clinical Trial Based on the Use of Mesenchymal Stem Cells From Autologous Bone Marrow in Patients With Lumbar Intervertebral Degenerative Disc Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Haematology Service,University Hospital of Salamanca, MªConsuelo del Cañizo Fernández-Roldán (Other); Spanish National Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSM/Fusión/2009
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Intervertebral Disc Disease
Keywords: Mesenchymal Stem Cells; Stem Cells; Intervertebral disc disease
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC seeded onto a phosphate ceramic (Experimental): Instrumented posterolateral fusion and autologous mesenchymal stem cells arranged in a phosphate ceramic.
  Interventions: Procedure: Instrumented posterolateral arthrodesis

INTERVENTIONS:
Procedure: Instrumented posterolateral arthrodesis — Cell suspension of mesenchymal stem cells (MSCs) obtained from bone marrow aspirate from the patient and expanded in vitro in a specific medium enriched with platelet lysate without addition of animal products.
  They used a minimum dose of 0.5 x106 CSM / kg and a maximum of 1, 5x106 CSM / kg of patient weight.
  Dosage Form: Suspension cell support hydroxyapatite and calcium phosphate Route of administration: placement in the fusion bed during surgery.

SUMMARY:
The purpose of this trial is to test the effectiveness of the use of a new therapeutic strategy in treating patients with degenerative disc disease lumbar intervertebral fusion with instrumented posterolateral autologous mesenchymal stem cells and arranged in a calcium phosphate ceramic (Conduit TM).

ELIGIBILITY:
Inclusion Criteria:

Clinical

* Box symptomatic (back pain and / or root) of lumbar degenerative disc disease monosegmental.
* Discopathy refractory to conservative treatment (drugs, physical therapy.)
* Evolution greater than or equal to 6 months. Radiological
* Discopathy radiation. Disc space narrowing, osteophytes, abnormal mobility, etc
* NMR: grades IV and V of Pfirman.

Exclusion Criteria:

* Rejection of surgical treatment.
* Systemic inflammatory disease (spondylitis, rheumatoid arthritis etc), tumor or infection.
* Immunosuppressive treatment.
* Congenital or acquired anatomical abnormality that prevents the surgical procedure.
* Neuropsychiatric pathology, drug addiction, psychosis, severe personality disorder.
* High surgical risk (ASA> IV), or contraindication to anesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-01; Primary Completion 2017-05-04 (Actual); Study Completion 2017-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Trauma Service. Hospital Universitario de Salamanca, Salamanca, Castille and León, Spain

REFERENCES:
- [Derived] Gomez-Ruiz V, Blanco JF, Villaron EM, Fidalgo H, Lopez-Parra M, Sanchez-Guijo F. Autologous mesenchymal stem cell transplantation for spinal fusion: 10 years follow-up of a phase I/II clinical trial. Stem Cell Res Ther. 2023 Apr 11;14(1):78. doi: 10.1186/s13287-023-03298-4. PMID 37038216
- [Derived] Blanco JF, Villaron EM, Pescador D, da Casa C, Gomez V, Redondo AM, Lopez-Villar O, Lopez-Parra M, Muntion S, Sanchez-Guijo F. Autologous mesenchymal stromal cells embedded in tricalcium phosphate for posterolateral spinal fusion: results of a prospective phase I/II clinical trial with long-term follow-up. Stem Cell Res Ther. 2019 Feb 22;10(1):63. doi: 10.1186/s13287-019-1166-4. PMID 30795797
- See also: Spanish cell therapy network (TerCel) — http://www.red-tercel.com
- See also: Salamanca University Foundation — http://fundacion.usal.es
- See also: Spanish Health Institute Carlos III — http://www.isciii.es